CLINICAL TRIAL: NCT02487095
Title: A Phase I/II Trial of Topotecan With VX-970 (M6620), an ATR Kinase Inhibitor in Small Cell Cancers
Brief Title: Trial of Topotecan With VX-970 (M6620), an ATR Kinase Inhibitor, in Small Cell Cancers and Extrapulmonary Small Cell Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Anish Thomas, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 150150; 15-C-0150
Record Dates: First submitted 2015-06-27; First posted 2015-07-01 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Carcinoma, Non-Small -Cell Lung; Ovarian Neoplasms; Small Cell Lung Carcinoma; Uterine Cervical Neoplasms; Carcinoma, Neuroendocrine; Extrapulmonary Small Cell Cancer
Keywords: RB1 Inactivation; Kinase Inhibitor; DNA Damage Response Network; MYC And CCNE1 Activation; Defective ATM-p53 Signaling Pathway
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Small Cell Lung Carcinoma; Uterine Cervical Neoplasms; Carcinoma, Neuroendocrine | interventions — Topotecan; berzosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Phase I VX-970 (M6620) + topotecan (Experimental): VX-970 (M6620) + topotecan at escalating doses
  Interventions: Drug: Topotecan; Drug: VX-970 (M6620)
- 2/Phase II VX-970 (M6620) + topotecan (Experimental): VX-970 (M6620) + topotecan at maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D)
  Interventions: Drug: Topotecan; Drug: VX-970 (M6620)

INTERVENTIONS:
Drug: Topotecan — Topotecan (in combination with VX-970 (M6620) administered by intravenous (IV) Days 1-5 in a 21 day cycle, until disease progression or development of intolerable side effects.
  Other Names: Hycamtin
Drug: VX-970 (M6620) — VX-970 (M6620 (in combination with Topotecan) administered by intravenous (IV) Day 5 or Days 2 and 5 in a 21 day cycle, until disease progression or development of intolerable side effects.
  Other Names: M6620

SUMMARY:
Background:

Chemotherapy damages cancer cell deoxyribonucleic acid (DNA) so the cells die, and the tumor shrinks. But it may stop working in some people over time. This is partly due to efficient DNA damage repair mechanisms used by tumor cells. VX-970 (M6620) may stop cancer cells from preventing the repair of DNA damaged by chemotherapy. The purpose of this study is to see if using the chemotherapy drug topotecan along with the drug VX-970 (M6620) will improve the response to chemotherapy.

Objective:

To study the safety and efficacy of VX-970 (M6620) and topotecan in treating small cell lung cancer.

Eligibility:

Adults at least 18 years old with small cell lung cancer.

Design:

Participants will be screened with medical history, physical exam, blood and heart tests, and scans. Most of these tests are part of their routine care. Most of these tests will be repeated throughout the study.

The study is set in 21-day cycles. Participants will get topotecan intravenous (IV) on days 1 through 5. They will get VX-970 (M6620) IV on day 5 alone or on day 5 and day 2.

Participants doctors will monitor them weekly for the first cycle, every 3 weeks after that.

For Part 1 of this Study the doses of topotecan and VX-970 (M6620) will be increased (according to the Protocol) to determine the maximum safe dose of the combination. The maximum safe dose of the combination is the dose at which no more than 1 in 6 people have an intolerable side effect.

More participants will join in Phase 2. They will take the drugs at the maximum safe dose, on the same schedule as the drugs were taken in Phase 1.

Participants will give samples of blood, hair, and tumor tissue (optional) at different times. They will discuss side effects at every visit.

A month after stopping taking the drugs, participants will have a physical exam and blood drawn. They will have follow-up phone calls every 3 months.

DETAILED DESCRIPTION:
Background:

Small cell lung cancer (SCLC) is an aggressive cancer with a poor prognosis.

Although highly responsive to chemotherapy initially, SCLC typically relapses quickly and becomes refractory to treatment within a few months.

There is only one Food and Drug Administration (FDA) approved treatment for patients with relapsed SCLC after first-line chemotherapy: topotecan, which inhibits religation of topoisomerase I-mediated single-strand deoxyribonucleic acid (DNA) breaks leading to lethal double-strand DNA breaks.

The survival of some SCLC cells despite initial tumor sensitivity to chemotherapy suggests the existence of a highly effective DNA damage response network.

SCLC is characterized by high replication stress (RB transcriptional corepressor 1 (RB1) inactivation, MYC and cyclin E1 (CCNE1) activation) and defective ataxia-telangiectasia mutated tumor protein p53 (ATM-p53) signaling pathway, which cause an excessive reliance on ataxia-telangiectasia rad 3-related (ATR) for survival following DNA damage.

We hypothesize that a combination of ATR kinase inhibition with DNA damaging agents such as topotecan will provide an attractive synthetically lethal therapeutic option for SCLC.

VX-970 is a potent and selective kinase inhibitor of ATR, and in vitro data support the hypothesis that ATR inhibition can improve SCLC responses to DNA damaging agents.

Primary objectives:

Phase 1: To identify the maximum tolerated dose (MTD) of topotecan in combination with VX-970.

Phase 2: To assess the efficacy with respect to clinical response rate of a combination of topotecan and VX-970 in the second-line treatment of patients with SCLC.

Eligibility:

Both Phase 1 and 2: Subjects must be greater than or equal to 18 years of age and have a performance status (Eastern Cooperative Oncology Group (ECOG) less than or equal to 2. Subjects must not have received chemotherapy or undergone major surgery within 4 weeks and radiotherapy within 24 hours prior to enrollment.

Phase 1: Subjects with histologically confirmed SCLC, non-small cell cancer (NSCLC), ovarian cancer, cervical cancer, and neuroendocrine cancers, and at least one prior chemotherapy. Patients with other histologies will be allowed if no standard treatment options exist. Patients with evaluable, but not measurable disease will be eligible for Phase I.

Phase 2: Subjects with histological confirmation of SCLC and one prior platinum-based chemotherapy. Patients with both platinum-sensitive and platinum-refractory disease will be eligible. Patients must have measurable disease to be eligible for Phase II.

Design:

Participants meeting inclusion and exclusion criteria will receive topotecan and VX-970 administered every 21 days (1 cycle), until disease progression or development of intolerable side effects.

Blood and hair samples will be collected at multiple time points during cycle 1 (pre-treatment on day 1, post treatment on days 2, and 3) for pharmacodynamic (PD) analyses.

Tumor biopsies, which are optional, will be obtained at baseline, during the first treatment cycle (approximately 15 hours after the first dose of VX-970 on day 3) and at disease progression except for subjects at the first dose level.

Participants at the first dose level will undergo biopsies on day 3 prior to third dose of topotecan.

Participants will be monitored weekly during the first cycle by clinic visit and basic labs.

Toxicity will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0, and tumor assessments will be made using computed tomography (CT) scans (chest, abdomen and pelvis) at baseline and after every 2 cycles according to Response Evaluation Criteria in Solid Tumors (RECIST) guideline version 1.1.

Follow-up for survival will be carried out every 3 months.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Both Phase I and Phase II:

  * Male and female subjects greater than or equal to 18 years of age. Because no dosing adverse event data are currently available on the use of topotecan in combination with VX-970 (M6620) in subjects less than 18 years of age, children are excluded from this study, but will be eligible for future pediatrics trials.
  * Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
  * Patients must have measurable disease, per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Subjects with evaluable, but not measurable disease will be eligible for Phase 1.
  * Subjects must not have received chemotherapy or undergone major surgery within 4 weeks and radiotherapy within 24 hours prior to enrollment.
  * Adequate organ functions

    * Hemoglobin greater than or equal to 9.0 g/dL
    * Absolute neutrophil count greater than or equal to 1.5x10^9/L
    * Platelets greater than or equal to 100x10^9/L
    * Total Bilirubin less than or equal to 2.0 mg/dL
    * Transaminases less than or equal to 2 x upper limit of normal (ULN) or if liver metastases were present, less than or equal to 3xULN
    * Creatinine less than or equal to 1.5 mg/dL or creatinine clearance by Cockcroft-Gault formula greater than or equal to 60 mL/min
  * Ability of subject to understand and the willingness to sign a written informed consent document.
  * The effects of VX-970 (M6620) on the developing human fetus are unknown For this reason and because topotecan is known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during study participation and for 6 months after the last dose study therapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Phase I:

  * Subjects with histologically confirmed small-cell lung cancer (SCLC), non- small cell lung cancer (NSCLC), ovarian cancer, cervical cancer, and neuroendocrine cancers will be eligible. Pathological confirmation of diagnosis will be done at National Cancer Institute (NCI) Laboratory of Pathology. Patients with other histologies will be allowed if no standard treatment options exist.
  * At least one prior chemotherapy
  * NSCLC subjects with epidermal growth factor receptor (EGFR) mutations or anaplastic lymphoma kinase (ALK) translocations should have previously received appropriate Food and Drug Administration (FDA) approved therapies in addition to prior chemotherapy
* Phase II:

  * Histological confirmation of SCLC, or extrapulmonary small cell cancer. Although NCI confirmation of pathology is not required prior to starting treatment, every effort will be made to obtain outside pathology to be reviewed by an NCI pathologist.
  * Subjects with both platinum-sensitive and platinum-refractory disease will be eligible

EXCLUSION CRITERIA:

* Subjects with tumor amenable to potentially curative therapy.
* Subjects who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to (study agent) or other agents used in study.
* Subjects with symptomatic brain metastases will be excluded from trial secondary to poor prognosis. However, subjects who have had treatment for their brain metastasis and whose brain disease is stable without steroid therapy for 1 week or on physiologic doses of steroids may be enrolled.
* Subjects requiring any medications or substances that are strong inhibitors or inducers of cytochrome p450, family 3, subfamily A (CYP3A) during the course of the study are ineligible. Lists including strong inhibitors and inducers of cytochrome p450 3A4 (CYP3A4) are provided.
* Subjects with evidence of severe or uncontrolled systemic disease, or any concurrent condition, which could compromise participation in the study, including, but not limited to, active or uncontrolled infection, immune deficiencies, Hepatitis B, Hepatitis C, uncontrolled diabetes, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, uncontrolled cardiac arrhythmia, stroke/cerebrovascular accident within the past 6 months, or psychiatric illness/social situations which would jeopardize compliance with the protocol.
* Human immunodeficiency virus (HIV)-positive subjects on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with VX-970 (M6620). In addition, these subjects are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Pregnant women are excluded from this study because topotecan is a Class D agent with the potential for teratogenic or abortifacient effects and because the effects of VX-970 (M6620) on the developing human fetus are currently unknown. In addition, because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with topotecan or VX-970 (M6620), breastfeeding should be discontinued if the mother is treated with these agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-07-30 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2024-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anish Thomas, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall AB, Newsome D, Wang Y, Boucher DM, Eustace B, Gu Y, Hare B, Johnson MA, Milton S, Murphy CE, Takemoto D, Tolman C, Wood M, Charlton P, Charrier JD, Furey B, Golec J, Reaper PM, Pollard JR. Potentiation of tumor responses to DNA damaging therapy by the selective ATR inhibitor VX-970. Oncotarget. 2014 Jul 30;5(14):5674-85. doi: 10.18632/oncotarget.2158. PMID 25010037
- [Background] Josse R, Martin SE, Guha R, Ormanoglu P, Pfister TD, Reaper PM, Barnes CS, Jones J, Charlton P, Pollard JR, Morris J, Doroshow JH, Pommier Y. ATR inhibitors VE-821 and VX-970 sensitize cancer cells to topoisomerase i inhibitors by disabling DNA replication initiation and fork elongation responses. Cancer Res. 2014 Dec 1;74(23):6968-79. doi: 10.1158/0008-5472.CAN-13-3369. Epub 2014 Sep 30. PMID 25269479
- [Background] Al-Ahmadie H, Iyer G, Hohl M, Asthana S, Inagaki A, Schultz N, Hanrahan AJ, Scott SN, Brannon AR, McDermott GC, Pirun M, Ostrovnaya I, Kim P, Socci ND, Viale A, Schwartz GK, Reuter V, Bochner BH, Rosenberg JE, Bajorin DF, Berger MF, Petrini JH, Solit DB, Taylor BS. Synthetic lethality in ATM-deficient RAD50-mutant tumors underlies outlier response to cancer therapy. Cancer Discov. 2014 Sep;4(9):1014-21. doi: 10.1158/2159-8290.CD-14-0380. Epub 2014 Jun 16. PMID 24934408
- [Result] Thomas A, Redon CE, Sciuto L, Padiernos E, Ji J, Lee MJ, Yuno A, Lee S, Zhang Y, Tran L, Yutzy W, Rajan A, Guha U, Chen H, Hassan R, Alewine CC, Szabo E, Bates SE, Kinders RJ, Steinberg SM, Doroshow JH, Aladjem MI, Trepel JB, Pommier Y. Phase I Study of ATR Inhibitor M6620 in Combination With Topotecan in Patients With Advanced Solid Tumors. J Clin Oncol. 2018 Jun 1;36(16):1594-1602. doi: 10.1200/JCO.2017.76.6915. Epub 2017 Dec 18. PMID 29252124
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-C-0150.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No participants were treated on Dose Level -1, Topotecan 1mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 105mg/m^2 IV on day 5.
Groups:
- Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5: Phase I Dose Level (DL) 1 Topotecan 1mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 140mg/m^2 IV on day 5
- Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5: Phase I Dose Level (DL) 2 Topotecan 1mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 140mg/m^2 IV on day 2, 5
- Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5: Phase I Dose Level (DL) 3 Topotecan 1.25mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 140mg/m^2 IV on day 2, 5
- Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5: Phase I Dose Level (DL) 4 Topotecan 1.25mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 210mg/m^2 IV on day 2, 5
- Phase II DL4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose: Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 210mg/m^2 IV on day 2, 5 Maximum Tolerated Dose/ Recommended Phase II Dose.
  26 participants with small cell lung cancer (SCLC) and 15 with extrapulmonary small cell cancer (EPSCC) are included in this Arm/Group.
Period: Phase I Dose Escalation
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 | Phase II DL4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose
Started | 6 | 6 | 3 | 6 | 0
Completed | 6 | 6 | 3 | 6 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 | Phase II DL4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose
Started | 0 | 0 | 0 | 0 | 41
Completed | 0 | 0 | 0 | 0 | 40
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Unable to scan/restage participant | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Phase II DL4 Topotecan 1.25mg/m^2 VX970 (M6620) 210mg/m^2 Recommended Phase II Dose: Phase I Dose Level (DL) 4 Topotecan 1.25mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 210mg/m^2 IV on day 2, 5 Maximum Tolerated Dose/Recommended Phase II Dose
  26 participants with small cell lung cancer (SCLC) and 15 with extrapulmonary small cell cancer (EPSCC) are included in this Arm/Group.
- Total: Total of all reporting groups
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 | Phase II DL4 Topotecan 1.25mg/m^2 VX970 (M6620) 210mg/m^2 Recommended Phase II Dose | Total
Number analyzed (Participants) | 6 | 6 | 3 | 6 | 41 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 3 | 5 | 28 | 47
  >=65 years | 0 | 1 | 0 | 1 | 13 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.98 (4.75) | 56.75 (15.43) | 57.17 (8.81) | 60.27 (5.73) | 59.67 (12.3) | 59.16 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 26 | 38
  Male | 3 | 3 | 0 | 3 | 15 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 5 | 6 | 3 | 6 | 38 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 5 | 6
  White | 6 | 4 | 3 | 6 | 35 | 54
  More than one race | 0 | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 3 | 6 | 41 | 62
Eastern Cooperative Oncology Group (ECOG) [Count of Participants; unit: Participants] — ECOG 0 is fully active. ECOG 1 is symptoms but ambulatory. ECOG 2 is in bed <50% of the time.
  Participants
    0 | 0 | 0 | 0 | 0 | 3 | 3
    1 | 6 | 6 | 3 | 6 | 38 | 59
    2 | 0 | 0 | 0 | 0 | 0 | 0
Tumor Type [Count of Participants; unit: Participants]
  Small-cell carcinoma | 1 | 1 | 0 | 3 | 26 | 31
  Mesothelioma | 2 | 1 | 1 | 1 | 0 | 5
  Non-small cell lung cancer | 1 | 1 | 0 | 0 | 0 | 2
  Pancreatic cancer | 0 | 1 | 1 | 0 | 0 | 2
  Rectal high-grade neuroendocrine carcinomas (HGNEC) | 0 | 1 | 0 | 1 | 0 | 2
  Cervical carcinoma | 1 | 0 | 0 | 0 | 0 | 1
  Ovarian cancer | 0 | 0 | 0 | 1 | 0 | 1
  Thymoma | 0 | 1 | 0 | 0 | 0 | 1
  Endometrial cancer | 1 | 0 | 0 | 0 | 0 | 1
  Cervical small-cell carcinoma | 0 | 0 | 1 | 0 | 3 | 4
  Small cell bladder vs prostate (tumor type undefined) | 0 | 0 | 0 | 0 | 1 | 1
  Small cell rectal | 0 | 0 | 0 | 0 | 1 | 1
  Small cell gallbladder | 0 | 0 | 0 | 0 | 1 | 1
  Small cell ovarian | 0 | 0 | 0 | 0 | 1 | 1
  Non-small cell lung cancer transformed to Small cell lung cancer | 0 | 0 | 0 | 0 | 3 | 3
  Small cell bladder cancer | 0 | 0 | 0 | 0 | 2 | 2
  Small cell breast cancer | 0 | 0 | 0 | 0 | 2 | 2
  Small cell prostate cancer | 0 | 0 | 0 | 0 | 1 | 1
Number of Participants That Received Prior Therapy [Count of Participants; unit: Participants] | 6 | 6 | 3 | 6 | 41 | 62

OUTCOME MEASURES:

1. Primary Outcome: Ph I: Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of Topotecan
Description: MTD is defined as the dose level at which no more than 1 of 6 subjects experience a dose-limiting toxicity (DLT) during one cycle of treatment. A DLT is defined using the Common Terminology Criteria in Adverse Events (CTCAE) v4.0 and is related or possibly drug related, such as neutropenia Grade 4 for >7 days duration, febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection), or Grade 3 thrombocytopenia. Death due to drug related adverse events.
Time Frame: End of Cycle 1, approximately 3 weeks
Measure: Number; unit: mg/m^2
Groups:
- All Participants: All participants in phase I DL1-DL4.
Arm/Group | All Participants
Number analyzed (Participants) | 21
mg/m^2 | 1.25

2. Primary Outcome: Ph I: Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) of VX-970 (M6620)
Description: as for outcome 1
Time Frame: End of Cycle 1, approximately 3 weeks
Measure: Number; unit: mg/m^2
Arm/Group | All Participants
Number analyzed (Participants) | 21
mg/m^2 | 210

3. Primary Outcome: Ph II: Number of Participants With a Clinical Response
Description: Clinical response was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete Response (CR) is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR) is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters. Progressive Disease (PD) is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). Stable Disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
Time Frame: Every two cycles (each cycle is 21 days) up to approximately 30 months.
Population: 1/26 participants was not evaluable for response in the Phase II DL4 SCLC group. Phase II, DL4 Arm/Group is split into two groups for this outcome measure because the distinction is relevant for the phase II, DL4 since extrapulmonary small cell cancers (EPSCC) was an exploratory cohort of the phase II DL4 (added with an amendment).
Measure: Count of Participants; unit: Participants
Groups:
- Phase II Dose Level 4 - Small Cell Lung Cancer (SCLC) Topotecan 1.25mg/m^2 IV/VX970 210mg/m^2 IV; Phase II DL 4 - Extrapulmonary Small Cell Cancer (EPSCC)Topotecan 1.25mg/m^2 IV/VX970 210mg/m^2 IV: Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 210mg/m^2 IV on day 2, 5.
  Maximum Tolerated Dose/Recommended Phase II Dose.
Arm/Group | Phase II Dose Level 4 - Small Cell Lung Cancer (SCLC) Topotecan 1.25mg/m^2 IV/VX970 210mg/m^2 IV | Phase II DL 4 - Extrapulmonary Small Cell Cancer (EPSCC)Topotecan 1.25mg/m^2 IV/VX970 210mg/m^2 IV
Number analyzed (Participants) | 25 | 15
Participants
  Complete Response | 0 | 0
  Partial Response | 9 | 3
  Progressive Disease | 2 | 6
  Stable Disease | 14 | 6

4. Primary Outcome: Number of Participants With Serious and Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 9 months and 9 days for Ph I DL1, 42 months and 12 days for Ph I DL2, 15 months and 9 days for Ph I DL3, 17 months and 9 days for Ph I DL4, and 43 months and 22 days for Ph II DL4.
Measure: Count of Participants; unit: Participants
Groups:
- Phase I DL 1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5: Phase I Dose Level (DL) 1 Topotecan 1mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 140mg/m^2 IV on day 5
- Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose: Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 210mg/m^2 IV on day 2, 5.
  Maximum Tolerated Dose/Recommended Phase II Dose.
  26 participants with small cell lung cancer (SCLC) and 15 with extrapulmonary small cell cancer (EPSCC) are included in this Arm/Group.
Arm/Group | Phase I DL 1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 | Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose
Number analyzed (Participants) | 6 | 6 | 3 | 6 | 41
Participants | 6 | 6 | 3 | 6 | 41

5. Secondary Outcome: Phase I: Progression-free Survival (PFS)
Description: PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first. Progression was assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) and is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study).
Time Frame: At disease progression - 0.68 months to 88.27 months, an Average Mean of 10.6 months
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5
Number analyzed (Participants) | 6 | 6 | 3 | 6
Months | 1.38 [0.85 to 35.56] | 7.88 [1.44 to 12.25] | 1.15 [0.85 to 14.88] | 5.025 [0.68 to 88.27]

6. Secondary Outcome: Phase II: Progression-free Survival (PFS)
Description: as for outcome 5
Time Frame: At disease progression, an average of 3.28 months.
Population: The Phase II, DL4 Arm/Group is split into two groups for this outcome measure because the distinction is relevant for the phase II, DL4 since extrapulmonary small cell cancers (EPSCC) was an exploratory cohort of the phase II DL4 (added with an amendment).1/26 participants was not evaluable for response in the Phase II DL4 SCLC group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase II Dose Level 4 - Small Cell Lung Cancer (SCLC) Topotecan 1.25mg/m^2 IV/VX970 210mg/m^2 IV | Phase II DL 4 - Extrapulmonary Small Cell Cancer (EPSCC)Topotecan 1.25mg/m^2 IV/VX970 210mg/m^2 IV
Number analyzed (Participants) | 25 | 15
Months | 4.6 [2.3 to 7.2] | 2.2 [0.9 to 2.9]

7. Secondary Outcome: Phase I and Phase II: Duration of Response (DOR)
Description: DOR is measured from the time measurement criteria are met for Complete Response (CR) or Partial Response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented in response to the combination in both platinum sensitive and refractory patients. CR is disappearance of all non-target lesions and normalization of tumor marker level. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: At disease progression, an average of 5.25 months.
Population: 1/26 participants were not evaluable in the Phase II DL4 SCLC group. The Phase II, DL4 Arm/Group is split into two groups for this outcome measure because the distinction is relevant for the phase II, DL4 since extrapulmonary small cell cancers (EPSCC) was an exploratory cohort of the phase II DL4 (added with an amendment). Only 1 participant was evaluable in Phase 1 DL1 and Phase 1 DL4.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase I DL 2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5: Phase I Dose Level (DL) 2 Topotecan 1mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 140mg/m^2 IV on day 2, 5
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL 2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 | Phase II Dose Level 4 - Small Cell Lung Cancer (SCLC) Topotecan 1.25mg/m^2 IV/VX970 210mg/m^2 IV | Phase II DL 4 - Extrapulmonary Small Cell Cancer (EPSCC)Topotecan 1.25mg/m^2 IV/VX970 210mg/m^2 IV
Number analyzed (Participants) | 1 | 6 | 3 | 1 | 25 | 15
Months | NA [66.5 to NA] — Median and Lower end of confidence interval is not estimable for 1 participant. | NA [NA to NA] — No partial response. | NA [NA to NA] — No partial response. | NA [53.4 to NA] — Median and Lower end of confidence interval is not estimable for 1 participant. | 4.9 [0.6 to 6.9] | 5.6 [4.4 to 6.9]

8. Secondary Outcome: Phase I: Overall Survival (OS)
Description: OS is defined as the time from the on-study date until date of death or last follow-up.
Time Frame: On-study date until date of death, an average of 17.65 months.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5
Number analyzed (Participants) | 6 | 6 | 3 | 6
Months | 5.125 [0.85 to 106.3] | 10.1 [2.3 to 42.3] | 3.844 [0.85 to 14.88] | 9.1 [3.84 to 94.84]

9. Secondary Outcome: Phase I: Number of Participants With a Change in H2AX Phosphorylation (ƴH2AX) Levels in Hairs From Baseline (Day 1 Pre-Treatment)
Description: Hair samples were obtained from participants to determine a change in H2AX phosphorylation (named ƴH2AX) in the hair follicles when compared to baseline (day 1 pre-treatment). ƴH2AX signals were detected by immunochemistry (microscopy) by using an antibody specific against ƴH2AX that, in turn, was detected by a secondary antibody conjugated to a fluorescent probe. ƴH2AX signal intensity was measured in bottom of hair bulbs.
  A change is defined as change in ƴH2AX signal (fluorescence intensity) in cells located toward the top of the hair bulbs.
Time Frame: Day 1 Pre-Treatment, Post treatment on day 2, and Post treatment on day 3
Population: 17/21 participants were analyzed in Phase I DL1 because these 17 patients had good quality hair samples (plucked hairs with good hair bulbs).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5
Number analyzed (Participants) | 5 | 4 | 3 | 5
Participants
  Post treatment on day 2 | 4 | 4 | 3 | 5
  Post treatment on day 3 | 5 | 4 | 3 | 5

10. Secondary Outcome: Phase I: Number of Participants With a Change in H2AX Phosphorylation (ƴH2AX) Levels in Peripheral Blood Mononuclear Cells (PBMCs) From Baseline (Day 1 Pre-Treatment)
Description: PBMCs were obtained from participants to determine a change in H2AX phosphorylation (named ƴH2AX) in peripheral blood mononuclear cells (PBMCs) when compared to baseline (day 1 pre-treatment). ƴH2AX was detected by immunochemistry (microscopy) by using an antibody specific against ƴH2AX that, in turn, was detected by a secondary antibody conjugated to a fluorescent probe. Changes in ƴH2AX levels in PBMCs is defined as changes in numbers of ƴH2AX foci per cells.
Time Frame: Day 1 Pre-Treatment, Post treatment on day 2, and Post treatment on day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5
Number analyzed (Participants) | 6 | 6 | 3 | 6
Participants
  Post treatment on day 2 | 5 | 2 | 3 | 3
  Post treatment on day 3 | 6 | 6 | 2 | 3

11. Secondary Outcome: Percentage of Peripheral Blood Mononuclear Cells (PBMCs): Cluster of Differentiation 14 (CD14)+ Monocytes Among Viable Cells, and Regulatory T Cells Among Cluster of Differentiation 4 (CD4)+ T Cells At Baseline and Post-Treatment
Description: Blood samples were collected via venipuncture and immunophenotyping of PBMCs were performed by multiparameter flow cytometry for CD14+ monocytes among viable cells, and regulatory T cells among CD4+ T cells.
Time Frame: Baseline and 3 weeks post-treatment
Population: Only one participant had a post treatment sample in phase 1 DL3.
Measure: Median (Inter-Quartile Range); unit: percentage of PBMCs
Groups:
- Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose: Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2 intravenous (IV) (days 1-5); VX970 (M6620) 210mg/m^2 IV on day 2, 5.
  Maximum Tolerated Dose/Recommended Phase II Dose.
  Small cell lung cancer (SCLC) participants only.
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 | Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose
Number analyzed (Participants) | 6 | 6 | 3 | 6 | 41
percentage of PBMCs
  Baseline CD14+ monocytes among viable cells | 33.30 [31.43 to 41.40] | 35.4 [22.10 to 46.83] | 38.20 [25.75 to 50.45] | 22.50 [18.05 to 36.93] | 34.25 [25.73 to 42.65]
  Post-Treatment CD14+ monocytes among viable cells: number analyzed (Participants) | 6 | 6 | 1 | 6 | 41
  Post-Treatment CD14+ monocytes among viable cells | 31.50 [29.45 to 34.18] | 34.95 [28.40 to 40.45] | 23.70 [NA to NA] — There was only 1 sample. | 33.25 [25.83 to 46.20] | 32.75 [27.80 to 47.85]
  Baseline regulatory T cells among CD4+ T cells | 3.19 [2.66 to 5.04] | 3.80 [2.66 to 4.18] | 3.32 [2.58 to 4.44] | 3.92 [3.14 to 4.30] | 3.50 [1.95 to 5.65]
  Post-Treatment regulatory T cells among CD4+ T cells: number analyzed (Participants) | 6 | 6 | 1 | 6 | 41
  Post-Treatment regulatory T cells among CD4+ T cells | 1.87 [1.78 to 3.04] | 4.42 [4.17 to 5.50] | 1.79 [NA to NA] — There was only 1 sample. | 3.11 [2.44 to 3.20] | 2.53 [1.68 to 3.37]

12. Secondary Outcome: Ratio of Peripheral Blood Mononuclear Cells (PBMCs): Cluster of Differentiation 8 (CD8)/Cluster of Differentiation 4 (CD4) T Cells at Baseline and Post-Treatment
Description: Blood samples were collected via venipuncture and immunophenotyping of PBMCs were performed by multiparameter flow cytometry for CD8/CD4 T cell ratio.
Time Frame: Baseline and 3 weeks post-treatment
Population: Only one participant had a post treatment sample in phase 1 DL3.
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL 2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 | Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose
Number analyzed (Participants) | 6 | 6 | 3 | 6 | 41
Ratio
  Baseline CD8/CD4 T cell ratio | 0.55 [0.48 to 0.96] | 1.12 [1.01 to 1.25] | 0.86 [0.64 to 0.87] | 1.10 [0.88 to 1.34] | 0.63 [0.36 to 0.97]
  Post treatment CD8/CD4 T cell ratio: number analyzed (Participants) | 6 | 6 | 1 | 6 | 41
  Post treatment CD8/CD4 T cell ratio | 0.64 [0.39 to 0.88] | 1.11 [0.88 to 1.26] | 0.29 [NA to NA] — There was only one sample. | 0.99 [0.54 to 1.41] | 0.58 [0.33 to 0.95]

13. Secondary Outcome: Phase II: Overall Survival (OS)
Description: OS is defined as the time from the on-study date until date of death or last follow-up.
Time Frame: On-study date until date of death, an average of 12.22 months.
Measure: Median (Full Range); unit: Months
Arm/Group | Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose
Number analyzed (Participants) | 41
Months | 6.5 [0.95 to 90.7]

14. Other Pre Specified Outcome: Phase I Number of Participants With a Dose Limiting Toxicity (DLT)
Description: A DLT is defined using the Common Terminology Criteria in Adverse Events (CTCAE) v4.0 and is related or possibly drug related, such as neutropenia Grade 4 for >7 days duration, febrile neutropenia (fever of unknown origin without clinically or microbiologically documented infection), or Grade 3 thrombocytopenia. Death due to drug related adverse events.
Time Frame: End of Cycle 1, approximately 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5
Number analyzed (Participants) | 6 | 6 | 3 | 6
Participants | 1 | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 9 months and 9 days for Ph I DL1, 42 months and 12 days for Ph I DL2, 15 months and 9 days for Ph I DL3, 17 months and 9 days for Ph I DL4, and 43 months and 22 days for Ph II DL4.
Arm/Group | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 | Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose
All-Cause Mortality (participants affected / at risk) | 5/6 | 6/6 | 3/3 | 5/6 | 35/41
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/6 | 3/3 | 5/6 | 25/41
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 3/3 | 6/6 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 (N=6) | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 (N=6) | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 (N=3) | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 (N=6) | Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose (N=41)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death NOS (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5)
Gastrointestinal disorders - Other, Black stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, altered mental status (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Coronavirus: Cough, lethargy, decreased oral intake, fever. (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Influenza-A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, Klebsiella bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Brain mets (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Death, Brain Mets (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Progressive disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Neutrophil count decreased (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, Liver ablation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, Liver embolization (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I DL1 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 5 (N=6) | Phase I DL2 Topotecan 1mg/m^2 Intravenous (IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 (N=6) | Phase I DL3 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 140mg/m^2 IV on Day 2, 5 (N=3) | Phase I DL4 Topotecan 1.25mg/m^2 Intravenous(IV) (Days 1-5); VX970 (M6620) 210mg/m^2 IV on Day 2, 5 (N=6) | Phase II Dose Level (DL) 4 Topotecan 1.25mg/m^2; VX970 (M6620) 210mg/m^2 Recommended Phase II Dose (N=41)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 13 (18)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 2 (4) | 0 (0) | 2 (2) | 6 (6)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (8) | 1 (1) | 2 (2) | 3 (4) | 22 (48)
Alkaline phosphatase increased (Investigations) | 1 (1) | 4 (11) | 2 (3) | 4 (5) | 29 (76)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 8 (8)
Anemia (Blood and lymphatic system disorders) | 6 (38) | 6 (78) | 3 (37) | 6 (53) | 39 (251)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (3) | 19 (30)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (7) | 2 (3) | 2 (4) | 3 (7) | 21 (50)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (6) | 0 (0) | 1 (2) | 6 (27)
Blurred vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
CPK increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 16 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 10 (11)
Creatinine increased (Investigations) | 1 (1) | 3 (4) | 1 (3) | 2 (3) | 15 (42)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (5)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 14 (24)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (9)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 10 (12)
Ear and labyrinth disorders - Other, Intermittent hearing impairment (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 8 (10)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Eye disorders - Other, Cornea scratched (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Decreased acuity left eye/wavy vision (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Miosis, Left side (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, Scotoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 11 (18)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (6) | 22 (31)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 2 (5) | 1 (1) | 0 (0) | 2 (3) | 8 (11)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Flu like symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Difficult Chewing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Port side erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Tingling sensation to legs and arms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, Tongue abrasion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gum infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 10 (14)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hepatic hemorrhage (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 8 (11)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3) | 1 (7) | 1 (2) | 2 (2) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (3) | 5 (6)
Hypernatremia (Metabolism and nutrition disorders) | 2 (7) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 2 (9) | 0 (0) | 0 (0) | 1 (3) | 5 (20)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (4) | 5 (28) | 3 (25) | 5 (23) | 30 (93)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 2 (5) | 2 (8) | 2 (12) | 21 (59)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 2 (4) | 2 (4) | 3 (9) | 3 (7) | 17 (43)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2) | 4 (16) | 1 (16) | 3 (8) | 16 (69)
Hyponatremia (Metabolism and nutrition disorders) | 3 (4) | 6 (61) | 3 (12) | 5 (33) | 30 (125)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 3 (10) | 2 (3) | 2 (6) | 23 (37)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (23)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Infections and infestations - Other, Zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, shingles (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 7 (8)
Infusion site extravasation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 6 (8)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localized edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Lymphocyte count decreased (Investigations) | 4 (42) | 6 (66) | 3 (14) | 6 (85) | 36 (267)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, Achilles tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (4)
Nausea (Gastrointestinal disorders) | 3 (4) | 5 (6) | 3 (4) | 2 (3) | 20 (40)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Other, Clonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, Hyperreflexia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, Loss sensation rectal/vagina (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, Myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, Paraneoplastic Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nervous system disorders - Other, R arm numbness and heaviness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (11) | 6 (18) | 2 (4) | 5 (13) | 22 (68)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5)
Otitis media (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 19 (29)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 6 (8)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Papilledema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 5 (11) | 5 (49) | 3 (9) | 5 (27) | 39 (193)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (5)
Psychiatric disorders - Other, Stress (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 9 (11)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Circular dermal eruptions (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Left arm rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Nodular lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Palpable subcutaneous nodules (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Penile derma eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Poison Ivy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Rash: R chest @ port site red/sore (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Skin lesions on dorsal hands (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Topical dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Skin and subcutaneous tissue disorders - Other, B/l leg rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Upper respiratory infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 17 (34)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Weight loss (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 17 (34)
White blood cell decreased (Investigations) | 5 (33) | 6 (33) | 3 (8) | 5 (24) | 30 (182)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/95/NCT02487095/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/95/NCT02487095/ICF_001.pdf